CLINICAL TRIAL: NCT03815708
Title: Heat Stress During Wheelchair Rugby and Basketball
Brief Title: Heat Stress in Wheelchair Sports
Status: Completed | Type: Observational
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2018-24
Record Dates: First submitted 2018-12-10; First posted 2019-01-24 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Heat Stress; Body Temperature Changes
MeSH Terms: conditions — Heat Stress Disorders; Body Temperature Changes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- wheelchair rugby players: well-trained spinal cord injured wheelchair rugby players
- wheelchair basketball players: well-trained spinal cord injured wheelchair basketball players

SUMMARY:
The aim of the study is to study the thermoregulatory responses under real life conditions, such as during wheelchair rugby and basketball matches. A further goal is to develop and validate a standardised field-based protocol, which induces the same thermoregulatory response as during a wheelchair rugby and basketball match. This knowledge allows to investigate strategies to reduce heat stress and to enhance exercise performance (e.g. pre-cooling) in the future, based on standardised conditions.

DETAILED DESCRIPTION:
A spinal cord injury leads to several physiological changes and complications, which might influence exercise performance (Perret and Abel, 2016). One major problem is the limited thermoregulation, especially in subjects suffering from a tetraplegia (Griggs et al., 2015; Price et al., 2006). There are only few studies, which investigated the thermoregulatory response during real life conditions in wheelchair athletes such as during a wheelchair rugby match (Griggs et al., 2017). However, to implement strategies to reduce heat stress (e.g. precooling methods) or to determine the influence of heat stress on exercise performance and to determine the effects of specific interventions the following two issues seem to be a prerequisite: First of all, we need to understand, which thermoregulatory response is induced under real life conditions, e.g. by a wheelchair rugby or basketball match. Second, if we want to study the effects of potential interventions, a standardised and reliable study protocol has to be available, which closely mimics match conditions and induces a similar amount of heat stress. Thus, the aim of the study is to measure thermoregulatory and physical performance outcomes during a real life wheelchair rugby and basketball match. A further goal is to develop and validate a standardised field-based protocol, which induces a similar thermoregulatory response as during a wheelchair rugby or basketball match. These knowledge builds the basis for future thermoregulatory studies based on a reliable and standardised field-based testing protocol.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature
* healthy, male or female wheelchair rugby (with tetraplegia) or basketball player (with paraplegia) of national or international level
* regularly taking part in competitions/games
* age between 18 and 60 years

Exclusion Criteria:

* asthma
* blood disorders
* actual injury, which impairs performance or other impossibility to exercise to exhaustion
* cardiovascular disease
* gastrointestinal disease, disorder or former surgery concerning the gastrointestinal tract
* not able to swallow a capsule
* less than 40kg of body mass
* MRI during the period of use of the e-Celsius® device

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: well trained spinal cord injured wheelchair rugby and basketball players
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Change in body core temperature | from 0 minutes to 32 minutes (cohort 1) or 48 minutes (cohort 2)
  recording body core temperature with an electronic capsule from the beginning to the end of a rugby or basketball game

SECONDARY OUTCOMES:
Change in heart rate | from 0 minutes to 32 minutes (cohort 1) or 48 minutes (cohort 2)
  heart rate from the beginning to the end of a rugby or basketball game
covered distance | 32 minutes (cohort 1) or 48 minutes (cohort 2)
  covered distance (meters) during a rugby or basketball game
Change in body weight | 32 minutes (cohort 1) or 48 minutes (cohort 2)
  difference in weight (kg) from before to after the game due to sweating and convection

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Perret, PD Dr., Principal Investigator — Swiss Paraplegic Centre, Guido A. Zäch Strasse 1, CH-6207 Nottwil
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No